CLINICAL TRIAL: NCT00860249
Title: Using Precision Performance Measurement To Conduct Focused Quality Improvement. Sub-study 2
Brief Title: Outreach for Patients That Are Newly Eligible for Colorectal Cancer Screening
Acronym: UPQUAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of sufficient participants meeting the eligibility criteria to complete study in proposed and acceptable time frame.
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kenzie Cameron, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HS017163-02 (AHRQ)
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2011-12-01 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-11

CONDITIONS: Colorectal Cancer
Keywords: education; preventive service; screening; Colorectal Cancer Screening; Prevention & Control
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): Usual Care. Participants in this arm will receive Usual care until outcome assessment is performed at 6 months following randomization. At that time, they will be sent a letter reminding them to obtain the ordered preventative service test, however no further outcomes will be assessed. Thus, during the course of the study, all participants in this arm will have solely received usual care.
- Behavioral: Letter Only (Experimental): Behavioral: Letter Only Prior to a scheduled upcoming appointment, participants will get a letter signed by their physician that provides brief information about colorectal cancer (CRC) and notes the importance of CRC screening.
  Interventions: Behavioral: Letter Only
- Behavioral: Letter and Educational DVD (Experimental): Behavioral: Letter and Educational DVD Participants will get a letter from their physician that provides brief information about colorectal cancer (CRC) and notes the importance of CRC screening. It will be accompanied by an educational DVD about the screening. The participants will receive this prior to a scheduled upcoming appointment with their physician.
  Interventions: Behavioral: Letter and Educational DVD

INTERVENTIONS:
Behavioral: Letter Only — Prior to a scheduled upcoming appointment, participants will get a letter signed by their physician that provides brief information about colorectal cancer (CRC) and notes the importance of CRC screening.
  Arms: Behavioral: Letter Only
Behavioral: Letter and Educational DVD — Participants will get a letter from their physician that provides brief information about colorectal cancer (CRC) and notes the importance of CRC screening. It will be accompanied by an educational DVD about the screening. The participants will receive this prior to a scheduled upcoming appointment with their physician.
  Arms: Behavioral: Letter and Educational DVD

SUMMARY:
The purpose of this study is to evaluate whether patient outreach is effective at increasing compliance with preventative screenings for those patients who, based on national quality standards, have become newly eligible for screening measures. We hypothesize that educational outreach may increase completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Northwestern Medical Faculty Foundation General Internal Medicine
* Patient has a scheduled appointment with a GIM physician in the next several weeks
* Patient will be 50 years old at the time of this appointment
* Patient is male or female

Exclusion Criteria:

* This is the first time the patient is seen in the NMFF GIM clinic
* There is a prior completion of CRC screening noted in EHR.
* There is a prior order placed for CRC screening in EHR.
* Patient has a history of CRC
* Patient has a diagnosis of ulcerative colitis, inflammatory bowel disease, Crohn's Disease, or documented colectomy.

Ages: 50 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Cameron, PhD, Principal Investigator — Northwestern University, Department of General Internal Medicine
Locations (1):
- Northwestern Medical Faculty Foundation General Internal Medicine Clinic, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial took place at a large urban academic primary care internal medicine practice in Chicago, IL. The trial enrolled patients between March and December 2009.
Pre-assignment Details: We used data contained in the clinic's electronic health record to identify eligible patients. All eligible patients were randomly assigned to one of the three study arms.
Groups:
- Usual Care: Usual Care. Participants in this arm will receive usual care until outcome assessment is performed at 6 months following randomization. At that time, they will be sent a letter reminding them to obtain the ordered preventative service test.
Period: Overall Study
Arm/Group | Usual Care | Behavioral: Letter Only | Behavioral: Letter and Educational DVD
Started | 21 | 18 | 21
Completed | 0 | 0 | 0
Not Completed | 21 | 18 | 21
Not completed — trial was terminated prior to completion | 21 | 18 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Behavioral: Letter Only | Behavioral: Letter and Educational DVD | Total
Number analyzed (Participants) | 21 | 18 | 21 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 21 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 14 | 42
  Male | 6 | 5 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 21 | 60

OUTCOME MEASURES:

1. Secondary Outcome: The Secondary Outcome for the Study is the Time to Screening Completion.
Description: This Outcome Measure would have reported the length of time, measured in days, that occurred between the date of randomization and the completed screening date. We planned to review the electronic health records of participants 6 months post randomization to look for either: (1)note in free text MD note documenting receipt of one form of CRC screening during study period or (2)lab results from fecal occult blood test, sigmoidoscopy, or colonoscopy. Screening completion equaled presence of a lab result or physician note in chart. No patient charts were reviewed due to low accrual.
Time Frame: 6 months after randomization
Population: Although 60 individuals were randomized to condition, the trial was halted prior to primary or secondary outcome chart reviews. Hence there are no results to report.
Measure: Number; unit: participants
Groups:
- Usual Care: Usual Care - participants receive usual care
- Behavioral: Letter Only: Participants in this arm will receive a letter signed by their physician that provides brief information about colorectal cancer (CRC) and notes the importance of CRC screening.
- Behavioral: Letter and Educational DVD: Participants will get a letter from their physician that provides brief information about colorectal cancer (CRC) and notes the importance of CRC screening. It will be accompanied by an educational DVD about the screening. The participants will receive this prior to a scheduled upcoming appointment with their physician.
Arm/Group | Usual Care | Behavioral: Letter Only | Behavioral: Letter and Educational DVD
Number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Usual Care vs Behavioral: Letter Only vs Behavioral: Letter and Educational DVD; Please note that no analyses were performed as the trial was stopped due to low enrollment; Test type: Superiority or Other; p < 0.017, Chi-squared — We used the Bonferroni calculation to adjust for the planned multiple comparisons among the three groups

2. Primary Outcome: Completion of CRC Screening
Description: What would have been reported as this Outcome Measure is the number of participants who completed screening. We planned to review electronic health records of participants 6 months post randomization to look for either: (1) note in free text MD note documenting receipt of one form of colorectal cancer (CRC) screening during study period or (2)lab results from fecal occult blood test, sigmoidoscopy, or colonoscopy. Screening completion equaled presence of a lab result or physician note in chart. No patient charts were reviewed due to low accrual.
Time Frame: 6 months from initial contact
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Usual Care | Behavioral: Letter Only | Behavioral: Letter and Educational DVD
Number analyzed (Participants) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Usual Care vs Behavioral: Letter Only vs Behavioral: Letter and Educational DVD; Please note that no analyses were performed as the trial was stopped due to low enrollment; Test type: Superiority or Other; p < 0.017, Chi-squared — We intended to use a Bonferroni calculation to adjust for multiple comparisons among study arms

ADVERSE EVENTS:
Arm/Group | Usual Care | Behavioral: Letter Only | Behavioral: Letter and Educational DVD
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18 | 0/21

LIMITATIONS AND CAVEATS:
Early termination prior to collection of primary or secondary outcome measures, hence no analyses of the primary or secondary outcomes were performed.Thus, the only results reported are baseline characteristics of enrolled participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes